CLINICAL TRIAL: NCT04519762
Title: Hupophosphatemia Levels Deleteriously Affect Outcome of Patients With Severe Sepsis/Septic Shock Admitted to ICU
Brief Title: Levels of 'Hypophosphatemia Affect Outcome of Septic Patients in ICU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Noha Sayed Hussien, Clinical Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: R38/2020
Record Dates: First submitted 2020-08-12; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Hypophosphatemia
MeSH Terms: conditions — Hypophosphatemia | interventions — alpha-glycerophosphoric acid; Sodium Chloride; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Management of sepsis/ septic shock via fluids, antibiotics, vasopressors and inotropes.
  Interventions: Drug: Antibiotics; Drug: Inotropes
- Study group (Active Comparator): Management of sepsis/ septic shock in addition to management of hypophosphatemia.
  Interventions: Drug: Glycophos (Sodium Glycerophosphate); Drug: Antibiotics; Drug: Inotropes

INTERVENTIONS:
Drug: Glycophos (Sodium Glycerophosphate) — Management of hypophosphatemia via Glycophos Management of severe sepsis/septic shock via fluid therapy, antibiotics, vasopressors and inotropics.
  Other Names: Saline
  Arms: Study group
Drug: Antibiotics — Management of severe sepsis/septic shock via fluid therapy, antibiotics, vasopressors and inotropics.
  Other Names: saline
Drug: Inotropes — Management of severe sepsis/septic shock via fluid therapy, antibiotics, vasopressors and inotropics.
  Other Names: saline

SUMMARY:
The current study aimed to determine the incidence of hypophosphatemia (HP) among severe sepsis/septic shock patients admitted to ICU and its impact on morbidity and mortality rates of these patients, and to evaluate the impact of phosphorous supplemental therapy (PST) on such outcomes.Thus, this study will hypothesize that diagnosis and management of HP may be advantageous for reduction of morbidity and mortality rates of septic patients admitted to ICU.

DETAILED DESCRIPTION:
The study will include all patients admitted to ICU with or developing severe sepsis or septic shock within 24-hr after admission to ICU. Patients will be categorized according to at-admission inorganic phosphate (Pi) level into normophosphatemia group and hypophosphatemia group (HP) (mild, moderate and severe HP). All patients will be evaluated using Sequential Organ Failure Assessment (SOFA) and Acute Physiology and Chronic Health Evaluation II score (APACHE II) and blood samples will be collected for ELISA estimation of serum Pi, human C-reactive protein (CRP), L-lactate, CBC picture , serum electrolytes and kidney and liver function tests. Serum Pi level will be re-estimated immediately and 24-hr after full dose administration. Outcomes will include the 28-day ICU morbidity and mortality rates and their relation to HP severity and PST administration.

Patients who will fulfill the inclusion criteria will be selectively divided into two groups according to estimated level of serum Pi: Control group will include patients with serum Pi >2.5 mg/dl and Study group will include patients having serum Pi<2.5 mg/dl and will be further sub-grouped according to severity of HP into mild HP (2-2.5 mg/dl), moderate (1-1.9 mg/dl) or severe (<1 mg/dl).

Central venous catheter will be inserted for all patients enrolled in the study via the jugular or subclavian vein. Then, baseline hemodynamic parameters and central venous pressure (CVP) will be estimated and will be continuously monitored. Arterial blood samples will be obtained anaerobically and collected in heparinized tubes for estimation of arterial blood gas and pH.

Sepsis management: Patients were managed according to guidelines of Surviving

Sepsis Campaign; briefly:

1. Fluid therapy
2. Vasoactive drug therapy
3. Intropics
4. Antibiotic therapy

HP management regimen follows:

1. Calculation of supplementation dose according to the equation: phosphate dose (in mmol) = 0.5 x body weight x (1.25 - [serum Pi]).
2. Preparation that will be used: Glycophos®, Fresenius Kabi Egypt (organic phosphate solution 1mmol/ml). Vial 20 ml (1ml contains 1mmol of phosphate and 2mmol of sodium).
3. Dilution: will be diluted prior to parenteral administration. 20 ml of sodium-glycerophosphate diluted in 30 cc of dextrose 5% administered by syringe pump (50 mL).
4. The total calculated dose will be divided into three doses every 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe sepsis and/or septic shock within 24 hours of admission to ICU

Exclusion Criteria:

* children and adulthoods younger than 18 years
* pregnancy
* severe hemorrhagic shock
* maintenance on immunosuppressant therapy for any indication
* patients who are expected to die within the first 24 hours after admission

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Mortality (No.) | 15 September 2020 - 15 December 2020 (3 months)
  Assessment of mortality Assessment of mortality
Mortality (%) | 15 September 2020 - 15 December 2020 (3 months)
  Assessment of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kamal, Dr., Principal Investigator — Ain Shams University

IPD SHARING:
Plan to Share IPD: No